CLINICAL TRIAL: NCT05598775
Title: Long-Term Safety Study of CTX0E03 in Subjects Who Completed PISCES III Study
Acronym: LTFU
Status: Enrolling by invitation | Type: Observational
Sponsor: ReNeuron Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: RN01-CP-0004
Record Dates: First submitted 2022-10-25; First posted 2022-10-28 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2022-10

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Other: Non Interventional long term safety follow up — Non Interventional long term safety follow up

SUMMARY:
The purpose of this long-term safety study is to follow up subjects treated with CTX0E03 DP to monitor for delayed oncological, neurological, and CTX0E03 DP-related adverse events and to monitor survival

DETAILED DESCRIPTION:
The goal of this study is to assess the long-term safety of subjects treated with intracerebral CTX0E03 DP as measured by the onset of delayed adverse events of special interest (AESIs). AESIs are defined as adverse events leading to death, new oncological adverse events, new neurological adverse events and any other adverse event, which in the opinion of the Safety/Project Physician is related to CTX0E03 DP.

ELIGIBILITY:
Inclusion Criteria:

Subjects who have received CTX0E03 DP as part of the active arm in the PISCES III study Have provided appropriate written informed consent

Exclusion Criteria:

* None

Ages: 35 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects who have received CTX0E03 DP as part of the active arm in the PISCES III study
Sampling Method: Non-Probability Sample
Enrollment: 9 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Long-term safety study is to follow up subjects treated with CTX0E03 DP | 4 Years
  Identify delayed oncological, neurological, and CTX0E03 DP-related adverse events and to monitor survival.

CONTACTS AND LOCATIONS:
Overall Officials: Amy Miller, RPh, PharmD, Principal Investigator — UBC
Locations (1):
- Amy Miller, RPh, PharmD, Morgantown, West Virginia, United States

IPD SHARING:
Plan to Share IPD: No